CLINICAL TRIAL: NCT01306513
Title: Effect of Autologous Bone Marrow Derived Mesenchymal Stromal Cells Prior to Lung Volume Reduction Surgery for Severe Pulmonary Emphysema- a Phase I Safety and Feasibility Study
Brief Title: Safety and Feasibility Study of Administration of Mesenchymal Stemcells for Treatment of Emphysema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Jan Stolk, MD PhD, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL28562.000.09
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Emphysema
Keywords: emphysema; lung volume reduction surgery; mesenchymal stromal cells
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cells (Experimental)
  Interventions: Biological: autologous bone marrow derived mesenchymal stromal cells

INTERVENTIONS:
Biological: autologous bone marrow derived mesenchymal stromal cells — Intravenous administration of autologous bone marrow-derived mesenchymal stromal cells.

SUMMARY:
The purpose of this study is to show safety and feasibility to administer patients own mesenchymal stem cells to show signs of repair of emphysematous lung tissue

DETAILED DESCRIPTION:
Study Rationale Emphysema is one of the two main components of chronic obstructive pulmonary disease (COPD) and contributes over many years to airway obstruction by the loss of elastic recoil around the smallest airways. Emphysema is induced by cigarette smoking and it is widely accepted that the disease is caused by excessive proteolytic activity by proteases and a chronic inflammatory process, characterized by a cellular influx consisting of macrophages, neutrophils and T cells. This inflammatory response is steroid resistant and leads to slow but persistent alveolar destruction, resulting in enlarged lungs with bullous parts in both lungs. In addition to a central role of innate immunity, recent studies suggest that also (auto)antigen specific immunity may play a role in the pathogenesis of COPD.

Currently, the only treatment available for severe emphysema is lung volume reduction surgery (LVRS) to remove the most destroyed parts of the lungs. The surgery is generally performed in two separate sessions with a 10-12 weeks interval, with each lung as a separate surgical target. This surgical treatment allows improved ventilation in the remaining less affected areas of the lungs as demonstrated by post-surgical clinical improvement of lung function and increased survival in a subgroup of patients. Delayed wound healing after LVRS is an important clinical problem. It may lead to prolonged hospital stay due to air leakage from the lungs into the thoracic cavity. Lung emphysema patients are at high risk for prolonged air leakage after this surgery, which is most likely explained by the inflammatory process related to the disease.

Mesenchymal stromal cells (MSC) are multipotent cells that can differentiate into several cell types, including fibroblasts, osteoblasts, adipocytes and chondrocyte progenitors. In recent years it has become evident that bone-marrow derived MSC (BM-MSC) have potent immunomodulatory effects on T and B cells and in animal models of chronic inflammation in vivo. In addition, it has been shown that MSC express or release a variety of soluble factors implicated in anti-apoptotic signaling and cell growth. Importantly, encouraging results have recently been obtained with the treatment of severe steroid resistant Graft versus Host Disease (GvHD) with donor (allogeneic) BM-MSC. Furthermore, in our institute autologous BM-MSC are currently under investigation for treatment of tissue injury due to autoimmune disease (Crohn's Disease) and allogeneic immune responses (renal transplant recipients with biopsy proven subclinical rejection). The combination of the immunosuppressive, growth-potentiating and anti-apoptotic properties of BM-MSC may lead to accelerated wound healing after LVRS and might induce lung repair. In the present phase I study the investigators will assess the safety and feasibility of intravenous (i.v.) administration of BM-MSC prior to LVRS in a small group of severe pulmonary emphysema patients. Results of this safety and feasibility study may lead to future studies on the use of BM-MSC for immunomodulation and induction of repair in patients with pulmonary emphysema and milder stages of COPD.

Objective To test the safety and feasibility of intravenous administration of autologous BM-MSC after one-sided LVRS and prior to a second LVRS procedure for patients with severe pulmonary emphysema.

Study design Open label, non-randomized, non-blinded, prospective clinical trial. Patients are operated in two sessions; initially on one lung without pre-surgical infusion of BM-MSC, followed by a second surgical procedure on the contralateral lung which is preceded by two i.v. infusions of BM-MSC one week apart, 4 and 3 weeks prior to the lung surgery.

Study population Patients of at least 40 years of age with end-stage emphysema who are eligible for lung volume reduction surgery.

Intervention The intervention consists of two doses of BM-MSC infusions in 10 patients with a one week interval, 4 and 3 weeks prior to the second LVRS respectively.

Study endpoints

Primary endpoint:

1. Safety and feasibility of intravenous infusion of two doses of BM-MSC with 1 wk interval after the first LVRS and prior to a second LVRS. Toxicity criteria will be evaluated by grade according to WHO.

Secondary endpoint:

1. Difference in days between post-surgical transpleural air leak of the lung in each patient after the first (no infusion of BM-MSC) and second surgical (3 weeks after the last i.v. infusion of BM-MSC) intervention.
2. Histological responses in resected lung tissue (measured by immunohistochemistry of markers of inflammation, fibrosis and repair).

ELIGIBILITY:
Inclusion Criteria:

* Class GOLD III for COPD

Exclusion Criteria:

* Patients with clinical and radiological evidence of bronchiectasis.
* Patients suffering from renal- or hepatic failure.
* A psychiatric, addictive, or any disorder that compromises ability to give truly informed consent for participation in this study.
* Use of any investigational drug within 1 month prior to screening.
* Patients with pulmonary hypertension, with mean PAP above 30 mmHg assessed by ultrasound of the chest or by transoesophageal ultrasound.
* Documented HIV infection.
* Active hepatitis B, hepatitis C or TB.
* Subjects who currently have or who have had an opportunistic infection (e.g., herpes zoster, cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, cardiac, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis).
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infra-clavicular, epitrochlear, or periaortic areas), or splenomegaly.
* Known recent substance abuse (drug or alcohol).
* Poor tolerability of venepuncture or lack of adequate venous access for required blood sampling during the study period.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
  Safety: rate and grade of (serious) adverse events in the study population using the WHO toxicity criteria. After infusion of MSC's investigators will score change in renal function, breathing rate, temperature, heart rate, and blood pressure.
  Feasibility: determination of the number of expanded MSCs in relation to the amount of autologous bone marrow collected, number of passages required and time to reach to study target dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stolk, MD, PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Department of Pulmonology, Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Stolk J, Broekman W, Mauad T, Zwaginga JJ, Roelofs H, Fibbe WE, Oostendorp J, Bajema I, Versteegh MI, Taube C, Hiemstra PS. A phase I study for intravenous autologous mesenchymal stromal cell administration to patients with severe emphysema. QJM. 2016 May;109(5):331-6. doi: 10.1093/qjmed/hcw001. Epub 2016 Jan 27. PMID 26819296